CLINICAL TRIAL: NCT03794765
Title: Use of Antibiotics as an Adjuvant in Patients With Acute Severe Ulcerative Colitis: A Randomised Trial
Brief Title: Antibiotics as an Adjuvant in Patients With Acute Severe Ulcerative Colitis
Acronym: AAASUC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vishal Sharma, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NK/5147/DM
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases; Acute Severe Colitis
Keywords: Antibiotics; Ceftriaxone; Metronidazole
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Ceftriaxone; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic (Experimental): Standard of Care (steroids, prophylactic anticoagulation, oral nutrition) And Antibiotics (Inj Ceftriaxone 1 gram intravenous twice daily And Inj Metronidazole 500 mg intravenous thrice daily) for initial 48 hours
  Interventions: Drug: Ceftriaxone; Drug: Metronidazole
- Placebo (Placebo Comparator): Standard of care (steroids, prophylactic anticoagulation, oral nutrition) And Placebo infusions similar to the active drugs
  Interventions: Other: Placebo infusion

INTERVENTIONS:
Drug: Ceftriaxone — Injection ceftriaxone 1 gm will be prepared by reconstitution of the crystallised powder form in 100 ml of normal saline. This preparation will then be infused slowly over thirty minutes, after intradermal testing for hypersensitivity. Inj ceftriaxone 1gm IV will be given twelve hourly.
  Arms: Antibiotic
Drug: Metronidazole — Injection metronidazole 500 mg is available from pharmacies in solutions of 100 ml. It will be infused slowly over thirty minutes, three times per day
  Arms: Antibiotic
Other: Placebo infusion — Similar placebo infusion
  Arms: Placebo

SUMMARY:
The study is planned as a randomised control trial to study the adjuvant use of antibiotics (ceftriaxone and metronidazole) to achieve a clinical response in hospitalised patients with acute severe ulcerative colitis

DETAILED DESCRIPTION:
All patients with active ulcerative colitis who present to the Outpatient department or the emergency services of PGIMER shall be screened. Those patients who have acute severe ulcerative colitis shall be assessed for inclusion into the study. Patients who fulfil the eligibility criteria will be randomised into two groups.

Group A will include patients in the intervention arm. They will be given intravenous antibiotics for three days. Injection ceftriaxone 1 gm will be prepared by reconstitution of the crystallized powder form in 100 ml of normal saline. This preparation will then be infused slowly over thirty minutes, after intradermal testing for hypersensitivity. Inj ceftriaxone 1gm IV will be given twelve hourly. Injection metronidazole 500 mg is available from pharmacies in solutions of 100 ml. It will be infused slowly over thirty minutes, three times per day, after intradermal testing for hypersensitivity. Both the drugs will be given for five days. In addition, they will receive the standard of care mentioned below.

Group B will include patients from the placebo arm. They will be given the standard of care as mentioned below. In addition, they will be infused 0.9 % saline of similar quantity, colour, and from similarly shaped bottles, for three days after sensitivity testing with the saline.

Detailed history and examination shall be done for all the patients. History regarding the stool output, any systemic symptoms, prior treatment history and history regarding any precipitant for the acute episode shall be taken. Examination will include vitals (pulse rate, blood pressure, temperature), general physical examination as well as an abdominal examination. All patients will undergo blood investigations on all three days. This includes a complete blood counts, kidney function tests, serum electrolytes, albumin, C-reactive protein, osteopontin, blood culture. Stool routine microscopic examination, fecal calprotectin, stool assay for clostridium difficile toxin will be done. X ray abdomen will be done on all three days to monitor the diameter of transverse colon. Patients will undergo an unprepared sigmoidoscopy with minimal air insufflation and mucosal biopsy. Biopsies will be taken for histological examination. Procalcitonin, fecal calprotectin and CRP shall be repeated on day 3 of admission.

All patients will be prescribed the standard treatment for acute severe colitis, which includes intravenous steroids (Inj Hydrocortisone 100 mg IV QID or Inj Methyprednisolone 60 mg iv OD), anticoagulation, (Inj Unfractionated heparin 5000 IU S/C BD), intravenous fluid supplementation and correction of electrolytes. Patients will be allowed orally and will be prescribed a diet of 25-30 kcal /kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Acute severe ulcerative colitis as described in European Crohn's and Colitis Organisation (ECCO) guidelines (adapted from Truelove and Witts)

Exclusion Criteria:

* Patients who deny consent
* Age<=12 years
* Pregnant or lactating women
* Severe uncontrolled comorbidities like diabetes mellitus, hypertension, coronary artery disease, chronic liver disease, chronic kidney disease, etc
* History of antibiotic use in the past one month, excluding those who may have received a single dose of antibiotic in past 24 hrs
* History of hypersensitivity or contraindication to steroids or the test drugs
* Presence of toxic megacolon as defined by transverse colon diameter more than 5.5cm on abdominal X-ray
* Patients with evidence of sepsis or active infection

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Clinical response as defined by the Oxford's criteria | 48 hours
  Patients will be defined as complete responders, partial responders or non-responders

SECONDARY OUTCOMES:
Proportion needing second line therapy | 28 days
  Second line therapy : Intravenous Infliximab, Intravenous cyclosporine or others
Proportion needing colectomy | 28 days
  Number of patients in each group needing colectomy
Mortality | 28 days
  Number of patients in having mortality
Duration of hospital stay | 28 days
  Length of hospital stay in each group
Change in serum CRP levels | 48 hours
Change in Mayo disease severity index | 48 hours
Patients with Reduction in fecal calprotectin by >100 mcg/mg | 48 hours
  Number of patients in each group having the predefined decline in fecal calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Sharma, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Shubhra Mishra, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mishra S, Mandavdhare HS, Singh H, Choudhury A, Shah J, Ram S, Kalsi D, Samanta J, Prasad KK, Sharma AK, Dutta U, Sharma V. Adjuvant use of combination of antibiotics in acute severe ulcerative colitis: A placebo controlled randomized trial. Expert Rev Anti Infect Ther. 2021 Jul;19(7):949-955. doi: 10.1080/14787210.2021.1856656. Epub 2020 Dec 14. PMID 33245002